CLINICAL TRIAL: NCT07013084
Title: Study on the Effect of Digital Smoking Cessation Education Intervention on Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: C202005128
Record Dates: First submitted 2025-05-26; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; virtual reality; outpatient
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D VR smoking cessation intervention (Experimental): The program consists of five sequential VR modules, each structured as an interactive game scenario targeting specific aspects of smoking behavior and cessation motivation.
  Interventions: Behavioral: 3D VR smoking cessation program
- comparison group (No Intervention): no 3D VR smoking cessation program intervention

INTERVENTIONS:
Behavioral: 3D VR smoking cessation program — Participants in the experimental group engaged with the VR system using a head-mounted display, allowing for full immersion in the virtual environment.
  Arms: 3D VR smoking cessation intervention

SUMMARY:
This study aimed to assess the novel approach of an immersive three-dimensional (3D) virtual reality (VR) smoking cessation program and its effectiveness on smoking outpatients

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) was conducted with 100 outpatients from a smoking cessation clinic in Taiwan. Participants were randomly assigned to either the experimental group (n=50) or the comparison group (n=50) through a coin toss. The experimental group received standard outpatient smoking cessation services in combination with an immersive 3D VR smoking cessation program, while the comparison group received only standard outpatient services. The VR program included five interactive modules that used immersive scenarios to simulate smoking-related cues and provide educational content, employing cognitive-behavioral techniques and practicing coping strategies to promote behavior change.

ELIGIBILITY:
Inclusion Criteria:

* currently receiving outpatient care at the smoking cessation clinic
* self-reported current tobacco use
* aged between 20 and 64 years
* no participation in any smoking cessation intervention within the past 12 months

Exclusion Criteria:

- Patients with medical contraindications that could prevent them from engaging with the VR equipment

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
smoking status indicator1 | From enrollment to the end of intervention at 12 weeks
  Participants reported the number of days they smoked in the past 30 days
smoking status indicator2 | From enrollment to the end of intervention at 12 weeks
  Participants reported the average number of cigarettes consumed per day in the past 30 days
smoking status indicator3 | From enrollment to the end of intervention at 12 weeks
  Nicotine dependence was measured using the FTND.
smoking status indicator4 | From enrollment to the end of intervention at 12 weeks
  exhaled CO levels were measured using a handheld CO monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital SongShan Branch ,Taipei,Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chun HR, Cheon E, Hwang JE. Systematic review of changed smoking behaviour, smoking cessation and psychological states of smokers according to cigarette type during the COVID-19 pandemic. BMJ Open. 2022 Jun 14;12(6):e055179. doi: 10.1136/bmjopen-2021-055179. PMID 35701057
- [Result] Keijsers M, Vega-Corredor MC, Tomintz M, Hoermann S. Virtual Reality Technology Use in Cigarette Craving and Smoking Interventions (I "Virtually" Quit): Systematic Review. J Med Internet Res. 2021 Sep 17;23(9):e24307. doi: 10.2196/24307. PMID 34533471
- [Result] Ebbert JO, Severson HH, Croghan IT, Danaher BG, Schroeder DR. Comparative effectiveness of the nicotine lozenge and tobacco-free snuff for smokeless tobacco reduction. Addict Behav. 2013 May;38(5):2140-5. doi: 10.1016/j.addbeh.2013.01.023. Epub 2013 Feb 4. PMID 23454876
- [Result] Tonnesen P, Lauri H, Perfekt R, Mann K, Batra A. Efficacy of a nicotine mouth spray in smoking cessation: a randomised, double-blind trial. Eur Respir J. 2012 Sep;40(3):548-54. doi: 10.1183/09031936.00155811. Epub 2012 Feb 9. PMID 22323576
- [Result] Caponnetto P, Cibella F, Mancuso S, Campagna D, Arcidiacono G, Polosa R. Effect of a nicotine-free inhalator as part of a smoking-cessation programme. Eur Respir J. 2011 Nov;38(5):1005-11. doi: 10.1183/09031936.00109610. Epub 2011 May 12. PMID 21565921
- [Result] Ward KD, Asfar T, Al Ali R, Rastam S, Weg MW, Eissenberg T, Maziak W. Randomized trial of the effectiveness of combined behavioral/pharmacological smoking cessation treatment in Syrian primary care clinics. Addiction. 2013 Feb;108(2):394-403. doi: 10.1111/j.1360-0443.2012.04048.x. Epub 2012 Nov 19. PMID 22882805
- [Result] Karekla M, Savvides SN, Gloster A. An Avatar-Led Intervention Promotes Smoking Cessation in Young Adults: A Pilot Randomized Clinical Trial. Ann Behav Med. 2020 Oct 1;54(10):747-760. doi: 10.1093/abm/kaaa013. PMID 32383736
- [Result] Goldenhersch E, Thrul J, Ungaretti J, Rosencovich N, Waitman C, Ceberio MR. Virtual Reality Smartphone-Based Intervention for Smoking Cessation: Pilot Randomized Controlled Trial on Initial Clinical Efficacy and Adherence. J Med Internet Res. 2020 Jul 29;22(7):e17571. doi: 10.2196/17571. PMID 32723722
- [Result] Pericot-Valverde I, Secades-Villa R, Gutierrez-Maldonado J. A randomized clinical trial of cue exposure treatment through virtual reality for smoking cessation. J Subst Abuse Treat. 2019 Jan;96:26-32. doi: 10.1016/j.jsat.2018.10.003. Epub 2018 Oct 16. PMID 30466545
- [Result] Guo JL, Liao JY, Chang LC, Wu HL, Huang CM. The effectiveness of an integrated multicomponent program for adolescent smoking cessation in Taiwan. Addict Behav. 2014 Oct;39(10):1491-9. doi: 10.1016/j.addbeh.2014.05.009. Epub 2014 May 28. PMID 24949950
- [Result] Borrelli B, Rueras N, Jurasic M. Delivery of a smoking cessation induction intervention via virtual reality headset during a dental cleaning. Transl Behav Med. 2021 Feb 11;11(1):182-188. doi: 10.1093/tbm/ibz144. PMID 31665495
- [Result] Giovancarli C, Malbos E, Baumstarck K, Parola N, Pelissier MF, Lancon C, Auquier P, Boyer L. Virtual reality cue exposure for the relapse prevention of tobacco consumption: a study protocol for a randomized controlled trial. Trials. 2016 Feb 19;17:96. doi: 10.1186/s13063-016-1224-5. PMID 26892001
- [Result] Park CB, Choi JS, Park SM, Lee JY, Jung HY, Seol JM, Hwang JY, Gwak AR, Kwon JS. Comparison of the effectiveness of virtual cue exposure therapy and cognitive behavioral therapy for nicotine dependence. Cyberpsychol Behav Soc Netw. 2014 Apr;17(4):262-7. doi: 10.1089/cyber.2013.0253. Epub 2014 Feb 20. PMID 24555521
- [Result] Bordnick PS, Traylor AC, Carter BL, Graap KM. A Feasibility Study of Virtual Reality-Based Coping Skills Training for Nicotine Dependence. Res Soc Work Pract. 2012 May;22(3):293-300. doi: 10.1177/1049731511426880. PMID 25484549
- [Result] Pericot-Valverde I, Garcia-Rodriguez O, Gutierrez-Maldonado J, Ferrer-Garcia M, Secades-Villa R. Evolution of smoking urge during exposure through virtual reality. Stud Health Technol Inform. 2011;167:74-9. PMID 21685645
- [Result] Gamito P, Oliveira J, Baptista A, Morais D, Lopes P, Rosa P, Santos N, Brito R. Eliciting nicotine craving with virtual smoking cues. Cyberpsychol Behav Soc Netw. 2014 Aug;17(8):556-61. doi: 10.1089/cyber.2013.0329. Epub 2014 Mar 24. PMID 24660864
- [Result] Acker J, MacKillop J. Behavioral economic analysis of cue-elicited craving for tobacco: a virtual reality study. Nicotine Tob Res. 2013 Aug;15(8):1409-16. doi: 10.1093/ntr/nts341. Epub 2013 Jan 15. PMID 23322768
- [Result] Garcia-Rodriguez O, Weidberg S, Gutierrez-Maldonado J, Secades-Villa R. Smoking a virtual cigarette increases craving among smokers. Addict Behav. 2013 Oct;38(10):2551-4. doi: 10.1016/j.addbeh.2013.05.007. Epub 2013 May 23. PMID 23793042
- [Result] Gamito P, Oliveira J, Baptista A, Morais D, Lopes P, Saraiva T, Rosa P, Santos N, Soares F, Sottomayor C, Barata F. Nicotine craving: ERPs correlates after VR exposure to smoking cues. Stud Health Technol Inform. 2012;181:78-82. PMID 22954832
- [Result] Ramon JM, Nerin I, Comino A, Pinet C, Abella F, Carreras JM, Banque M, Baena A, Morchon S, Jimenez-Muro A, Marqueta A, Vilarasau A, Bullon R, Masuet-Aumatell C. A multicentre randomized trial of combined individual and telephone counselling for smoking cessation. Prev Med. 2013 Sep;57(3):183-8. doi: 10.1016/j.ypmed.2013.05.014. Epub 2013 Jun 1. PMID 23732247
- [Result] Free C, Knight R, Robertson S, Whittaker R, Edwards P, Zhou W, Rodgers A, Cairns J, Kenward MG, Roberts I. Smoking cessation support delivered via mobile phone text messaging (txt2stop): a single-blind, randomised trial. Lancet. 2011 Jul 2;378(9785):49-55. doi: 10.1016/S0140-6736(11)60701-0. PMID 21722952
- [Result] Morris CD, Waxmonsky JA, May MG, Tinkelman DG, Dickinson M, Giese AA. Smoking reduction for persons with mental illnesses: 6-month results from community-based interventions. Community Ment Health J. 2011 Dec;47(6):694-702. doi: 10.1007/s10597-011-9411-z. Epub 2011 May 10. PMID 21556784
- [Result] Reitzel LR, McClure JB, Cofta-Woerpel L, Mazas CA, Cao Y, Cinciripini PM, Vidrine JI, Li Y, Wetter DW. The efficacy of computer-delivered treatment for smoking cessation. Cancer Epidemiol Biomarkers Prev. 2011 Jul;20(7):1555-7. doi: 10.1158/1055-9965.EPI-11-0390. Epub 2011 May 25. PMID 21613389